CLINICAL TRIAL: NCT07355816
Title: Effect of Different Root Canal Disinfection Procedures on Postoperative Pain: A One-Week Follow-Up Clinical Study
Brief Title: Effect of Different Root Canal Disinfection Procedures on Postoperative Pain
Acronym: EDRCD-PP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, İbrahim AKDENİZ, Specialist dentist / Endodontist, Cumhuriyet University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2022-11/01
Record Dates: First submitted 2025-11-19; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Pain, Postoperative
Keywords: Root Canal Therapy,Disinfection Methods
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- conventional needle irrigation (Experimental): Conventional needle irrigation(CNI) Group: A total of 6 mL of 2.5% NaOCl was delivered in three cycles using a 31-gauge irrigation needle positioned 2 mm short of the working length. Each cycle lasted 20 seconds, followed by a 20-second waiting period. Subsequently, 2 mL of 17% Ethylenediaminetetraacetic acid(EDTA) (Imicryl Dental, Konya, Türkiye) was applied for 1 minute, followed by another 1-minute waiting period, and finally 2 mL of distilled water was used as the final rinse.
  Interventions: Procedure: Conventional Needle Irrigation
- Passive Ultrasonic Irrigation Group (Experimental): Passive ultrasonic irrigation(PUI) Group: Passive ultrasonic activation was performed with an ultrasonic device (Ultra X, Eighteeth, Changzhou, China) using a 20/.02 tip during the waiting periods used in the CNI group. The ultrasonic tip was positioned 2 mm short of the working length and activated vertically with 2-3 mm strokes without contacting the canal walls.
  Interventions: Procedure: Passive Ultrasonic Irrigation
- Sonic Irrigation Group (Experimental): Sonic irrigation(SI) Group: Sonic activation was performed using a polymer tip (Dentsply Tulsa Dental Specialties) loosely fitted into the canal and placed 2 mm short of the working length during the waiting periods used in the CNI group. The tip was activated by vertical in-and-out motion to induce sonic agitation.
  Interventions: Procedure: Sonic Irrigation
- KTP Laser Disinfection Group (Experimental): Potassium titanyl phosphate(KTP) Laser Group: In this group, after shaping was completed, the final irrigation procedure was carried out as in the CNI group. Following irrigation, the root canals were dried with sterile paper points at the working length. Then, KTP laser irradiation (SMARLITE D, DEKA laser system, Calenzano FI, Italy) was applied in a pulsed mode at 1.5 W power (Ton: 20 ms, Toff: 50 ms). A 200 µm fiber tip attached to the handpiece was inserted 1 mm short of the working length and moved coronally in a spiral motion for 5 seconds. After each 5-second irradiation, a 20-second interval was allowed, and the process was repeated five times. Laser safety protocols were strictly followed, and protective goggles were used by the operator, assistant, and patient.
  Interventions: Procedure: KTP Laser Disinfection

INTERVENTIONS:
Procedure: Conventional Needle Irrigation — Root canals will be irrigated using a conventional syringe and needle technique with standard irrigant solutions. This method relies solely on manual delivery without activation devices.
  Arms: conventional needle irrigation
Procedure: Passive Ultrasonic Irrigation — Root canals will be irrigated using passive ultrasonic activation, which uses ultrasonic energy to improve irrigant effectiveness and reduce microbial load beyond manual techniques.
  Arms: Passive Ultrasonic Irrigation Group
Procedure: Sonic Irrigation — Root canals will be irrigated using a sonic activation device (e.g., EndoActivator) to enhance irrigant penetration and bacterial elimination compared to conventional irrigation.
  Arms: Sonic Irrigation Group
Procedure: KTP Laser Disinfection — Root canals will be disinfected using a KTP laser following standard irrigation protocols. Laser application aims to provide enhanced antimicrobial effects not achievable with conventional or activated irrigation methods.
  Arms: KTP Laser Disinfection Group

SUMMARY:
This clinical study evaluated the effects of different root canal disinfection procedures on postoperative pain. Patients requiring root canal treatment received one of several disinfection methods. Postoperative pain was assessed at 6,24, 48, 72 hours and on the 7th day using a standard pain scale. The aim of the study was to identify which method resulted in the least discomfort. Participation involved a single treatment session and short-term follow-up for pain measurement.

ELIGIBILITY:
Inclusion criteria

* Systemically healthy individuals between the ages of 18 and 65,
* Adequate mouth opening,
* Asymptomatic devitaled mandibular premolar with a single root and single canal,
* Negative response to cold and electric pulp tests and no bleeding at the pulp chamber opening,
* Able to provide rubber dam isolation,
* Presence of opposing teeth.

Exclusion criteria

* Presence of mental or psychiatric disorders,
* Allergic diseases,
* Use of painkillers within 12 hours or antibiotics within 1 week before the procedure,
* Swelling, palpation/percussion pain, or sinus tract before treatment,
* Presence of a periodontal pocket greater than 3 mm in diameter on the involved tooth,
* Presence of a periapical radiolucency greater than 5 mm in diameter associated with the involved tooth,
* Initiation of root canal treatment,
* Irreparable material loss, root fracture, or crack,
* Severe mobility,
* Open apex,
* Severe root canal calcification,
* Internal or external resorption,
* Bruxism,
* Complaints of pain elsewhere in the mouth or in a tooth,
* Being pregnant or breastfeeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-06-13 (Actual); Primary Completion 2024-11-11 (Actual); Study Completion 2024-11-11 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain Intensity | 6, 12, 24, 48, and 72 hours after root canal treatment
  Postoperative pain intensity assessed using the Visual Analog Scale (VAS), ranging from 0 to 100, where 0 indicates no pain and 100 indicates the worst pain imaginable; higher scores indicate greater pain severity

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cumhuriyet University, Sivas, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2022-12-15): https://cdn.clinicaltrials.gov/large-docs/16/NCT07355816/Prot_ICF_000.pdf